CLINICAL TRIAL: NCT06481150
Title: A Novel Approach for Reducing Hyperoxaluria and Kidney Stone Risk.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jonathan Whittamore, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU-2023-1257; 1UL1TR003163 (NIH)
Record Dates: First submitted 2024-06-24; First posted 2024-07-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria | interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tenapanor (Experimental): 30 mg Tenapanor twice a day
  Interventions: Drug: Tenapanor
- Placebo (Placebo Comparator): 30 mg Placebo twice a day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tenapanor — Each tablet 30 mg
  Other Names: XPHOZAH; IBSRELA
  Arms: Tenapanor
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This pilot study is proposing a novel approach to directly target intestinal oxalate absorption with the drug Tenapanor, which was recently FDA-approved for treating hyperphosphatemia in patients with chronic kidney disease. Tenapanor works by blocking paracellular phosphate absorption by the intestine, but the underlying mechanisms have not been clearly defined. Since phosphate and oxalate ions are absorbed through the same paracellular pathway, and are of similar size and charge, Tenapanor is hypothesized to also reduce dietary oxalate absorption and consequently lower urinary oxalate excretion.

DETAILED DESCRIPTION:
The proposed proof-of-concept studies will determine whether Tenapanor reduces urine oxalate in normal human subjects receiving a high-oxalate diet in a crossover placebo-controlled short-term metabolic study.

Study Design Screening - One 24-hour urine for analysis of stone-risk profile, one blood sample for comprehensive metabolic panel and cystatin C, one stool sample for fecal calprotectin, physical exam, social and medical history, vital signs, demographic information, personal information.This is a two-phase study, each phase is 5 days in duration.

Phase 1: The subjects will consume a pre-prepared oxalate-rich metabolic diet for 5 days while taking 30 mg Tenapanor or Placebo twice a day just prior to the morning and evening meals. On days 4 and 5 they will collect two 24-hour urines for measurement of urine oxalate and stone-risk profile.

Washout: The subjects will undergo a 9-day washout period. Phase 2: The subjects will consume a pre-prepared oxalate-rich metabolic diet for 5 days while taking 30 mg Tenapanor or Placebo twice a day just prior to the morning and evening meals. On days 4 and 5 they will collect two 24-hour urines for measurement of urine oxalate and stone-risk profile.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy adult volunteers

Exclusion Criteria:

* Personal history of kidney stones
* Pregnant or nursing
* Recurrent urinary tract infections
* Lithogenic urine chemistry at baseline (oxalate > 45 mg/24 h, urine calcium > 300 mg/24 h)
* Chronic kidney disease (eGFR < 90 mL/min/1.73m2)
* Personal history of GI disease, GI obstruction, or GI surgery
* Chronic diarrhea
* Intestinal inflammation (Fecal calprotectin > 120 mcg/g)
* Drugs which are substrates of OATP2B1 (e.g. enalapril)
* Chronic use of sodium polystyrene sulfonate, angiotensin-converting enzyme inhibitors, diuretics, antacids, alkali treatment, or carbonic anhydrase inhibitors.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-14 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
24-h urine oxalate | Two 24-h urine on days 4 and 5 of each arm
  Study participants collect two 24-hour urine specimens for analysis of their stone-risk profile, including oxalate (mg/24 h), comparing placebo with drug treatment (Tenapanor).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Whittamore, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King AJ, Siegel M, He Y, Nie B, Wang J, Koo-McCoy S, Minassian NA, Jafri Q, Pan D, Kohler J, Kumaraswamy P, Kozuka K, Lewis JG, Dragoli D, Rosenbaum DP, O'Neill D, Plain A, Greasley PJ, Jonsson-Rylander AC, Karlsson D, Behrendt M, Stromstedt M, Ryden-Bergsten T, Knopfel T, Pastor Arroyo EM, Hernando N, Marks J, Donowitz M, Wagner CA, Alexander RT, Caldwell JS. Inhibition of sodium/hydrogen exchanger 3 in the gastrointestinal tract by tenapanor reduces paracellular phosphate permeability. Sci Transl Med. 2018 Aug 29;10(456):eaam6474. doi: 10.1126/scitranslmed.aam6474. PMID 30158152

DOCUMENTS (1):
  • Informed Consent Form (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT06481150/ICF_000.pdf